CLINICAL TRIAL: NCT02119832
Title: A Prospective Clinical Evaluation of the TVA FLEX-1 Device Protocol Flex-1-002-IR Intervention Reduction
Brief Title: A Prospective Clinical Evaluation of the Total Vascular Access (TVA) FLEX-1 Device Protocol Flex-1-002-IR Intervention Reduction (IR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLEX-1-002-IR
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Chronic kidney disease; Arteriovenous fistula; Hemodialysis; Vascular access
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endovascular AVF (EndoAVF) (Experimental): The FLEX System will be used to endovascularly create a fistula in CKD patients who require hemodialysis vascular access
  Interventions: Device: Endovasccular AVF (EndoAVF)

INTERVENTIONS:
Device: Endovasccular AVF (EndoAVF) — The FLEX System will be used to endovascularly create a fistula in CKD patients who require hemodialysis vascular access
  Other Names: FLEX

SUMMARY:
The primary objective of this clinical study is to evaluate the preliminary safety and effectiveness of using the FLEX-1 device for the creation of an arteriovenous fistula (AVF) including coiling of the brachial vein during the index procedure in patients requiring chronic hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for a native surgical arteriovenous fistula, as determined by the treating physician.
* Adult (age >18 years old).
* Advanced chronic kidney disease (CKD), stage 4 or 5 electing for hemodialysis.
* Written informed consent obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  The safety of the FLEX-1 system based on the overall complication rates derived from adverse event data.

SECONDARY OUTCOMES:
Access Functionality | 6 months
  The functionality of the AVF will be measured based on use of the AVF with two needles for at least 75% of dialysis sessions over a 4-week period following at least a one month maturation period.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Italian Hosptial, Asuncion, Paraguay
Locations (1):
- Italian Hospital, Asunción, Paraguay